CLINICAL TRIAL: NCT00514774
Title: Ursodiol in Huntington's Disease
Acronym: UDCA-HD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: Huntington Study Group (Network); Huntington Society of Canada (Other)
Responsible Party: Penelope Hogarth, MD, Oregon Health & Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00001927
Record Dates: First submitted 2007-08-08; First posted 2007-08-10 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Huntington Disease
Keywords: Huntington chorea; chorea; hereditary; tauroursodeoxycholic acid; ursodeoxycholic acid; TUDCA; UDCA
MeSH Terms: conditions — Huntington Disease; Chorea | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental)
  Interventions: Drug: ursodiol
- B (Experimental)
  Interventions: Drug: ursodiol
- C (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ursodiol — ursodiol 300 mg twice daily for study days 0 through 28
  ursodiol 600mg twice daily on study days 0 through 28
  Other Names: Ursodeoxycholic acid; UDCA
  Arms: A; B
Drug: placebo — placebo 600mg twice daily for study days 0 through 28
  Arms: C

SUMMARY:
The purpose of this study is to evaluate the safety of the drug ursodiol (ursodeoxycholic acid, UDCA) in people with Huntington's disease (HD) and to explore how the compound is processed by the body.

DETAILED DESCRIPTION:
Huntington's disease is an inherited neurodegenerative disease that causes a movement disorder, dementia, and psychiatric and behavioral disturbance in affected individuals.

Tauroursodeoxycholic acid (TUDCA) is a bile acid synthesized in the liver by the conjugation of taurine to ursodeoxycholic acid (UDCA). It is thought to function as an anti-apoptotic agent in HD, evidenced by studies in toxic cell models and both toxic and transgenic rodent models of the disease.

Ursodiol is a commercially-available exogenous form of UDCA, the precursor of TUDCA. Although the compound has an established dosing, safety, tolerability and efficacy profile in patients with hepatobiliary disorders, gaps exist in the understanding of the pharmacokinetics / pharmacodynamics of the compound, particularly in patients with normal gastrointestinal function, and no human data exist for its therapeutic use in neurodegenerative disorders. The specific aims of this study are:

1. To establish whether treatment with the drug ursodiol will result in measurable levels of its bile acid metabolites in serum and CSF at standard oral doses; and whether a dose-response can be detected using these measures.
2. To establish a preliminary safety and tolerability profile of the drug in subjects with HD.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will be age 18 or older
* All subjects will have manifest Huntington disease determined by clinical exam plus either documented prior DNA testing for the HD gene or a documented family history of the disease

Exclusion Criteria:

* Subjects taking oral contraceptives, cholestyramine, colestipol, or aluminum-based antacids will be excluded
* Subjects with known allergy or other contraindication to the study drug will be excluded
* Subjects with bleeding diathesis, or on coumadin or mandatory aspirin will be excluded
* Subjects with unstable medical or psychiatric illness will be excluded
* Subjects with clinically significant lab / EKG abnormalities at screening will be excluded
* Subjects who are currently pregnant or breastfeeding will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Safety measures (complete blood count, chemistry profile, electrocardiogram, urinalysis) | 35 days
Tolerability measures (adverse event severity) | 35 days
Pharmacokinetic measures (Serum and CSF levels of bile acids) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Penelope Hogarth, M.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Keene CD, Rodrigues CM, Eich T, Chhabra MS, Steer CJ, Low WC. Tauroursodeoxycholic acid, a bile acid, is neuroprotective in a transgenic animal model of Huntington's disease. Proc Natl Acad Sci U S A. 2002 Aug 6;99(16):10671-6. doi: 10.1073/pnas.162362299. Epub 2002 Jul 29. PMID 12149470
- [Background] Keene CD, Rodrigues CM, Eich T, Linehan-Stieers C, Abt A, Kren BT, Steer CJ, Low WC. A bile acid protects against motor and cognitive deficits and reduces striatal degeneration in the 3-nitropropionic acid model of Huntington's disease. Exp Neurol. 2001 Oct;171(2):351-60. doi: 10.1006/exnr.2001.7755. PMID 11573988
- See also: Official website for the Huntington Study Group — http://www.huntington-study-group.org/